CLINICAL TRIAL: NCT06000475
Title: Enhancing Memory in Cognitive Processing Therapy for Older Adults With PTSD
Brief Title: Enhancing Memory in CPT for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: D4627-P; 1I21RX004627 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Psychotherapy; Memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded to treatment status during feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Processing Therapy (CPT) (Active Comparator): Standard CPT as described in the treatment manual
  Interventions: Behavioral: Cognitive Processing Therapy
- Cognitive Processing Therapy (CPT) + Memory Support (Experimental): CPT+Memory support will also incorporate frequent and intentional use of strategies to enhance learning and memory of this content.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Cognitive Processing Therapy (CPT) + Memory Support

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT as described in the treatment manual
  Other Names: CPT
Behavioral: Cognitive Processing Therapy (CPT) + Memory Support — CPT+Memory support will also incorporate frequent and intentional use of strategies to enhance learning and memory of this content.
  Arms: Cognitive Processing Therapy (CPT) + Memory Support

SUMMARY:
Several psychotherapies for posttraumatic stress disorder (PTSD) have a strong evidence base for their efficacy, but nonresponse rates are high, particularly among older Veterans. Accumulating evidence indicates that memory deficits and poor learning of therapy contents adversely affect psychotherapy treatment response in PTSD. However, limited research has examined methods for increasing learning of therapy contents in psychotherapy for PTSD. The proposed study aims to examine the feasibility of integrating an intervention to increase learning and memory of psychotherapy content into the provision of a widely used psychotherapy, cognitive processing therapy (CPT), for older adults with PTSD. The ultimate goal of this line of research is to develop novel rehabilitation interventions to increase functioning for individuals with PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is prevalent among Veterans and is a substantial public health burden. Several psychotherapies, including cognitive processing therapy (CPT), have a strong evidence base for their efficacy in PTSD. However, many individuals show limited benefit from such treatments, particularly older Veterans. One factor likely affecting treatment response is poor encoding, storage, and retrieval of the skills and treatment points that are learned in psychotherapy. Individuals with PTSD display deficits in learning and memory, and aging is independently associated with declines in memory and executive functioning. Thus, older adults with PTSD may be at heightened risk of cognitive dysfunction that could impact their ability to benefit from frontline PTSD treatments. To this end, pre-treatment memory functioning has been shown to consistently predict treatment response in psychotherapy for PTSD. Inefficient learning and memory for psychotherapy content may be one mechanism explaining this relationship, as poor learning of therapy content is linked with worse treatment adherence and outcomes. The primary aim of this proposal is to examine the feasibility and acceptability of integrating a novel Memory Support intervention into the provision of CPT for older adults with PTSD. The Memory Support intervention was developed such that specific strategies to enhance encoding and retrieval of therapy content and skills can be integrated into manualized psychotherapy. However, no prior studies have integrated this intervention into treatments for PTSD. The proposed project will be guided by a user-centered design framework for treatment development and be conducted in three phases. In the first phase, the investigators will develop a modified CPT treatment manual that systematically integrates Memory Support, with clinician (n=3) and Veteran (n=3) feedback to provide guidance on process and techniques. In the next phase, the investigators will conduct iterative refinement of the modified treatment through a case series in older Veterans (n=3) with an experienced CPT therapist. Finally, the investigators will conduct a small feasibility randomized controlled trial (n=20) in which the investigators will examine accrual, retention, completion, acceptability, and variability in symptom and functional outcomes, as well as all procedures for a larger trial. The proposed project offers substantial conceptual innovations by bridging foundational work from rehabilitation neuropsychology and psychotherapy mechanisms research and will provide valuable pilot data to inform a novel intervention for older Veterans with PTSD that can be tested in future large-scale studies. Such approaches may be especially relevant for Veterans with neurocognitive deficits (e.g., memory), potentially suggesting a target for a personalized approach to mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with DSM-5 diagnoses of PTSD via the Clinician Administered PTSD Scale (CAPS-5)
* Age >59

Exclusion Criteria:

* daily benzodiazepine use (due to memory impairing effects)
* bipolar or psychotic disorders
* current suicidal ideation with plan or intent
* current moderate or severe substance use disorder not in remission for >1 mo.
* severe traumatic brain injury
* a Montreal Cognitive Assessment (MoCA) indicative of dementia
* or other disorders that would severely limit study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist-5 (PCL-5) | Through study completion, weeks 12-16 of treatment
  Questionnaire for symptoms of PTSD; the range of the scale is from 0 (no symptoms) to 80 (maximal symptoms).

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | Through study completion, weeks 12-16 of treatment
  8-item patient satisfaction scale; the range of the scale is from 8 to 32, where low scores are indicative of low satisfaction and high scores are indicative of high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Scott, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No